CLINICAL TRIAL: NCT03181854
Title: Randomized Controlled Trial of Integrated Early Palliative Care for Advanced Cancer Patients
Brief Title: Randomized Controlled Trial of Integrated Early Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Evidence-Based Healthcare Collaborating Agency (Other Government); National Institute of Health, Korea (Other Government); National Clinical Research Coordination Center, Seoul, Korea (Other Government); Seoul National University Bundang Hospital (Other); Severance Hospital (Other); Gyeongsang National University Hospital (Other); Chungnam National University Hospital (Other); Chonbuk National University Hospital (Other); Daegu Fatima Hospital (Other); Hallym University Medical Center (Other); Korea University Guro Hospital (Other); Asan Medical Center (Other); Chonnam National University Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Pohang Semyeong Christianity Hospital (Unknown); Gangneung Asan Hospital (Other)
Responsible Party: Principal Investigator, Young Ho Yun, Principal Investigator, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HC15C1391-1
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Advanced Cancer; Solid Tumor
Keywords: Integrated Early Palliative Care
MeSH Terms: interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Consultation with PCT doctor every 3 weeks. Telephone coaching once a week for 3 months and once in 2 weeks for another 3 months.
  Interventions: Behavioral: Telephone coaching; Behavioral: Consultation with PCT doctor
- Control Group (No Intervention): Usual palliative care can be provided if desired.

INTERVENTIONS:
Behavioral: Telephone coaching — Telephone coaching about overcoming the crisis is provided once a week for 3 months and once in 2 weeks for another 3 months.
  Arms: Intervention group
Behavioral: Consultation with PCT doctor — Consultation with PCT physician every 3 weeks.
  Arms: Intervention group

SUMMARY:
This study verifies whether integrated Early Palliative Care for advanced cancer patients diagnosed due to a solid tumor improve quality of life and enhances the ability to overcome the current crisis.

DETAILED DESCRIPTION:
Previous reports suggest that starting palliative care early in cancer patients appears to improve patient's quality of life, symptom management, depression, and anxiety.

This study aims to evaluate the effect of the introduction of early palliative care services to advanced cancer patients. Eligible patients are 20 years or older, and has an advanced cancer diagnosis (histologically or cytologically confirmed) due to a solid tumor, a European Cooperative Oncology Group performance status of 0-2, an estimated life expectancy of 12 months or less. The primary goal of an integrated early palliative care program is to improve the overall quality of life of patients and their families. Secondarily, it is to help understand the disease, resolving conflicts in the decision-making process, improving the crisis coping capacity, and further determining the patient's and family's advanced care planning. At last, it is desired to evaluate the effect of the program on overall medical cost savings and 1 year survival.

Participants of the study will be allocated in the intervention group and the control group equally. Within three weeks from the time of randomization, the first meeting with a palliative care team will be held. In the time of baseline questionnaire, patients will be provided with self-study education materials and videos on the early palliative care and advance care planning. Once in every three weeks for six months, which is the duration for one treatment course, palliative care for advance care planning, symptom control, and other mental, social and spiritual problems will be provided. After the first meeting with the palliative care team, telephone coaching will be performed once a week for the first 12 weeks and then every two weeks until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject 20 years and older.
* Subject who has an advanced cancer diagnosis (histologically or cytologically confirmed) due to a solid tumor
* Subject whose ECOG performance status is between 0 to 2.
* Subject with an estimated life expectancy of 12 months and less (assessed by the treating oncologist)
* Subject who volunteers

Exclusion Criteria:

* Inability to speak, understand or write Korean.
* Medical conditions that would limit adherence to participation of the clinical trial(as confirmed by their referring physician; e.g. dyspnea)
* Suspension of all cancer treatment
* Palliative care consultation at any time or in palliative care

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in level of EORTC QLQ-C15-PAL | baseline, 12 weeks, 18 weeks, 24 weeks
  A questionnaire developed to assess the quality of life of palliative cancer care patients.

SECONDARY OUTCOMES:
Change in level of MQOL | Baseline, 12 weeks, 18 weeks, 24 weeks
  A questionnaire that measures psychological, existential well-being, and support.
Change in level of EQ-5D of EuroQoL | Baseline, 12 weeks, 18 weeks, 24 weeks
  A questionnaire that measures mobility, self-care, daily activity, pain/discomfort, and anxiety/depression.
Change in level of PHQ-9 | Baseline, 12 weeks, 18 weeks, 24 weeks
  9-question instrument given to patients in a primary care setting to screen for the presence and severity of depression.
Change in level of Understanding the illness | Baseline, 12 weeks, 18 weeks, 24 weeks
  2 questions to assess how patients understand the prognosis of their illness
Change in level of Crisis Overcoming Capability(SAT-SF) | Baseline, 12 weeks, 18 weeks, 24 weeks
  A questionnaire about goal of life, current crisis/goal, positivity, preparation and practice.
Change in Advance Care Preference | Baseline, 12 weeks, 18 weeks, 24 weeks
  Questions about advance directive and treatment preference in case of terminal condition
Medical cost and utilization of CAM | 12 weeks, 24 weeks
  Overall medical cost savings (cost effectiveness) and use of complementary and alternative medicine
1 year survival | 1 year
  1 year survival
Changes of CQOL | Baseline, 12 weeks, 18 weeks, 24 weeks
  A questionnaire that measures quality of life and burden for family caregivers
Change in level of PHQ-9 of family caregivers | Baseline, 12 weeks, 18 weeks, 24 weeks
  9-question instrument given to caregivers in a primary care setting to screen for the presence and severity of depression.
Change in level of Understanding the illness of family caregivers | Baseline, 12 weeks, 18 weeks, 24 weeks
  2 questions to assess how family caregivers understand the prognosis of patients' illness
Change in level of Crisis Overcoming Capability(SAT-SF) of family caregivers | Baseline, 12 weeks, 18 weeks, 24 weeks
  A questionnaire about goal of life, current crisis/goal, positivity, preparation and practice of family caregivers.
Change in Advance Care Preference of family caregivers | Baseline, 12 weeks, 18 weeks, 24 weeks
  Questions about family caregivers' preference on advance directive and treatment in case of terminal condition
Change in Quality Care Questionnaire | Baseline, 12 weeks, 3 months after death
  The 4-factor, 32-item Quality Care Questionnaire-Palliative Care (QCQ-PC), which covers appropriate communication with health care professionals (ten items), discussing value of life and goals of care (nine items), support and counseling for needs of holistic care (seven items), and accessibility and sustainability of care (six items).

CONTACTS AND LOCATIONS:
Overall Officials: Young Ho Yun, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (10):
- South Korea (10):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jung JY, Yun JY, Kang JH, Koh SJ, Kim YJ, Seo S, Kim JH, Cheon J, Kang EJ, Song EK, Nam EM, Oh HS, Choi HJ, Kwon JH, Bae WK, Lee JE, Jung KH, Kang E, Yun YH. Interaction effect of comorbid depression and proactive positivity coping strategy on the 1-year survival of patients with advanced cancer: a nationwide multicentre study in South Korea. BMC Psychiatry. 2025 Jun 2;25(1):565. doi: 10.1186/s12888-025-06972-4. PMID 40457290
- [Derived] Kang E, Kang JH, Koh SJ, Kim YJ, Seo S, Kim JH, Cheon J, Kang EJ, Song EK, Nam EM, Oh HS, Choi HJ, Kwon JH, Bae WK, Lee JE, Jung KH, Yun YH. Early Integrated Palliative Care in Patients With Advanced Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2024 Aug 1;7(8):e2426304. doi: 10.1001/jamanetworkopen.2024.26304. PMID 39115845